CLINICAL TRIAL: NCT07307560
Title: High-Flow Nasal Cannula for Preventing Hypoxia During Sedated Endoscopy in High-Risk Obstructive Sleep Apnea Patients: A Multicenter Randomized Trial
Brief Title: High-Flow Nasal Cannula for Preventing Hypoxia During Sedated Endoscopy in High-Risk Obstructive Sleep Apnea Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chief Physician,Researcher, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZJU2025C207
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hypoxia; Esophageal Cancer; Gastric Cancer (Diagnosis); Obstructive Sleep Apnea (OSA)
Keywords: Sedation; Hypoxia; Obstructive Sleep Apnea (OSA); Gastrointestinal Endoscopy
MeSH Terms: conditions — Hypoxia; Esophageal Neoplasms; Stomach Neoplasms; Disease; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal cannula Group (Experimental): In this group, patients use the High-flow nasal cannula
  Interventions: Device: High-flow nasal cannula Group
- Regular Nasal Cannula Group (Active Comparator): In this group, patients use the regular nasal cannula for oxygenation.
  Interventions: Device: Regular Nasal Cannula

INTERVENTIONS:
Device: High-flow nasal cannula Group — Using High-flow nasal cannula oxygenation
  Arms: High-flow nasal cannula Group
Device: Regular Nasal Cannula — Using regular nasal cannula for oxygenation
  Arms: Regular Nasal Cannula Group

SUMMARY:
Hypoxia represents the most frequent adverse event during propofol-sedated gastrointestinal endoscopy. The STOP-BANG questionnaire serves as a widely adopted, straightforward tool for screening obstructive sleep apnea (OSA) risk, with a score ≥5 identifying high-risk OSA patients who are particularly susceptible to hypoxia under sedation. Although preliminary research from our team suggests that High-Flow Nasal Cannula (HFNC) may lower the incidence of hypoxemia, evidence remains limited and inconsistent in studies specifically targeting high-risk OSA populations. Therefore, this multicenter randomized controlled trial aims to evaluate whether HFNC can effectively reduce the occurrence of hypoxia during sedated gastrointestinal endoscopy in patients identified as high-risk for OSA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* STOP-Bang score ≥5.
* Scheduled for sedated gastrointestinal endoscopy (gastroscopy, colonoscopy, or combined gastroscopy + colonoscopy).
* The estimated duration of the procedure does not exceed 45 minutes.
* Patients have signed the informed consent form.

Exclusion Criteria:

* Coagulation disorders or bleeding tendency (e.g., oral/nasal bleeding risk, mucosal injury, space-occupying obstructions).
* Active upper respiratory tract infection (oral, nasal, or pharyngeal), or fever (core temperature >37.5°C).
* Chronic obstructive pulmonary disease or other acute/chronic pulmonary diseases requiring long-term or intermittent oxygen therapy, or preoperative SpO₂ ≤ 92% on room air.
* Severe organ dysfunction, including: Cardiac insufficiency (<4 METs), Severe renal insufficiency (requiring dialysis), Diagnosed severe hepatic insufficiency, Increased intracranial pressure, ASA physical status ≥ IV.
* Confirmed pregnancy or current breastfeeding.
* Known allergy to sedatives (e.g., propofol) or medical adhesives.
* Multiple traumatic injuries.
* Current participation in another clinical trial.
* Other conditions deemed unsuitable by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-12-21 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  75% ≤ SpO2 < 90% for <60 s

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  90% ≤ SpO2 < 95%
The incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s

OTHER OUTCOMES:
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Hospital Of Jiaxing, Jiaxing, Zhejiang
  - Quzhou People's Hospital, Quzhou, Zhejiang